CLINICAL TRIAL: NCT00387673
Title: Effect of Prolonged Electrical Stimulation on Neural Plasticity in SCI
Brief Title: Effect of Prolonged Electrical Stimulation on Neural Plasticity in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B4439-R
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-05

CONDITIONS: Spinal Cord Injury
Keywords: electrical stimulation; hand; Rehabilitation; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): 6 weeks of upper extremity training for 3 sessions/week, as follows: a) somatosensory stimulation of the median, ulnar and radial nerves at the level of the wrist (2 hours/session);
  Interventions: Behavioral: Somatosensory Stimulation and Massed Practice Training
- Arm 2 (Active Comparator): a 6-week period of 2 hours somatosensory stimulation of the hand, without training
  Interventions: Behavioral: Somatosensory Stimulation and Massed Practice Training
- Arm 3 (Placebo Comparator): a 6-week period of 2 hours sham somatosensory stimulation of the hand, followed by 1 hour of activity-based training
  Interventions: Behavioral: Somatosensory Stimulation and Massed Practice Training

INTERVENTIONS:
Behavioral: Somatosensory Stimulation and Massed Practice Training — a) somatosensory stimulation of the median, ulnar and radial nerves at the level of the wrist (2 hours/session); SS group b) somatosensory stimulation of the median, ulnar and radial nerves at the wrist (2 hours/session) followed by an activity-based upper extremity training program (1 hour/session); SS+ABT group and c) sham somatosensory stimulation of the median, ulnar and radial nerves at the wrist (2 hours/session) followed by an activity-based upper extremity training program (1 hour/session); ABT group then carry out training in the 3 subject groups simultaneously, each group consisting of 2 subjects at a time, with 2 sets of subjects/year over a 2-year period, yielding a target sample of 36 subjects.

SUMMARY:
Electrical stimulation (pulses of electricity applied over the skin of your wrist) and activity-based hand exercise have been shown to improve motor skill and strength in individuals with stroke and have recently been shown to also have an effect on individuals with spinal cord injury. Therefore, the purpose of this research study is to investigate whether electrical stimulation alone or electrical stimulation followed by activity-based training produces gains in pinch strength (how hard you can squeeze your thumb and pointer finger together) and upper extremity function (how well your arm and hand can perform activities) in individuals with spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) affects 10,000 individuals per year in the United States. Approximately one half of all individuals with SCI have tetraparesis due to cervical injury. Impaired hand function significantly limits the ability of individuals with cervical SCI to perform manual activities of daily living which affects these individuals physically, psychologically and socially. Preliminary research by this investigator suggests that somatosensory stimulation combined with activity-based training improves hand function and strength in individuals with incomplete cervical SCI. Further investigations on these novel techniques are warranted due to the need to establish proven effective rehabilitation techniques that promote recovery of function in individuals with SCI.

The purpose of this research study is to: 1)determine if somatosensory stimulation in the form of prolonged, peripheral nerve electrical stimulation can enhance the effect of an upper extremity activity-based training program in individuals with incomplete cervical SCI, and if so, 2) identify the operative neural mechanisms underlying the changes induced with the application of somatosensory stimulation.

The hypotheses of this study are that individuals with incomplete cervical SCI:

1. a 6-week period of somatosensory stimulation of the hand, either alone or combined with activity-based training, will produce improvements in behavioral outcomes that are significantly greater than those produced by activity-based training preceded by a sham stimulation period
2. this behavioral improvement will be associated with greater changes in cortical excitation than will be observed in subjects receiving activity-based training preceded by a sham stimulation period.

The specific objectives of this study are to:

1. Recruit male and female volunteers with spastic paresis due to incomplete SCI with impaired hand function, and randomize subjects into 1 of 3 groups, each of which receives 6 weeks of upper extremity training for 3 sessions/week, as follows: a) somatosensory stimulation of the median, ulnar and radial nerves at the level of the wrist (2 hours/session); SS group b) somatosensory stimulation of the median, ulnar and radial nerves at the wrist (2 hours/session) followed by an activity-based upper extremity training program (1 hour/session); SS+ABT group and c) sham somatosensory stimulation of the median, ulnar and radial nerves at the wrist (2 hours/session) followed by an activity-based upper extremity training program (1 hour/session); ABT group then carry out training in the 3 subject groups simultaneously, each group consisting of 2 subjects at a time, with 2 sets of subjects/year over a 2-year period, yielding a target sample of 36 subjects.
2. Conduct pre-and post-training assessments of behavioral outcomes using Wolf Motor Function Test and Jebsen Taylor Hand Function test to measure upper extremity function, hand-held dynamometry to measure pinch grip strength, and Semmes-Weinstein Monofilament Testing to measure sensory function.
3. Conduct pre-and post-training assessments of supraspinal motor recruitment, including motor evoked potential (MEP) amplitudes in response to transcranial magnetic stimulation and extent and duration of cortical silent period in response to transcranial magnetic stimulation; and spinal motoneuron excitability measured by F-wave amplitude and persistence.

ELIGIBILITY:
Inclusion Criteria:

* Trace voluntary thumb movement or able to pick up small objects with a tenodesis grip
* Between ages 18 and 60
* Spastic paresis (manifest as spasms, clonus, and/or hyperreflexia) due to neurologically incomplete SCI
* Medically stable
* Communicate questions/needs and answer yes/no questions reliably.

Exclusion Criteria:

* Altered cognitive status
* Level of injury caudal to the C7 level
* History of CVA, seizures
* Implanted metal devices in the head, less than one year post injury, and severe spasticity of the muscles of the upper extremities (defined by a score of 2 or higher on the Modified Ashworth Spasticity Scale)
* Patients with pacemakers will also be excluded from this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Medical Center, Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 0 (Project has officially closed. PI for this project has left VA without forwarding information) | 0 (Project has officially closed. PI for this project has left VA without forwarding information) | 0 (Project has officially closed. PI for this project has left VA without forwarding information)
Completed | 0 (Project has officially closed. PI for this project has left VA without forwarding information) | 0 (Project has officially closed. PI for this project has left VA without forwarding information) | 0 (Project has officially closed. PI for this project has left VA without forwarding information)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Project has officially closed. PI for this project has left VA without forwarding information.
Arm/Group | Effect of Prolonged Electrical Stimulation on Neural Plastici
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
  Female | 0
  Male | 0
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Conduct pre-and Post-training Assessments of Behavioral Outcomes Using Wolf Motor Function Test and Jebsen Taylor Hand Function Test to Measure Upper Extremity Function, Hand-held Dynamometry to Measure Pinch Grip Strength, and Semmes-Weinstein Monofilam
Time Frame: Outcome measures: baseline, 6 weeks after baseline, post testing, 6 weeks post testing
Population: Project has officially closed. PI for this project has left VA without forwarding information.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Project has officially closed. PI for this project has left VA without forwarding information.
Arm/Group | Project Closed
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No